CLINICAL TRIAL: NCT05599204
Title: Effect Of Schroth Method On Balance In Upper Crossed Syndrome
Acronym: UCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam omran Grase, principle investigator mariam omran grase, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003993
Record Dates: First submitted 2022-10-19; First posted 2022-10-31 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Postural; Defect
Keywords: Schroth Method; upper cross syndrome; balance
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus

STUDY DESIGN:
Intervention Model Description: Schroth exercise and postural correction group
Who Masked: Investigator, Outcomes Assessor
Masking Description: opaque sealed envelop
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- schroth exercise (Experimental): the patients will receive Schroth exercise twice a week for four weeks
  Interventions: Other: schroth exercise; Other: postural correction exercise
- postural correction exercise (Active Comparator): the patients will receive postural correction exercise twice a week for four weeks
  Interventions: Other: postural correction exercise

INTERVENTIONS:
Other: schroth exercise — the patients will receive the Schroth three-dimensional exercise. patient first assumes a posture in the cervico-cranial and shoulder girdle and the thoracic region is held in the correct posture. The patient inspires air into the concave side and during the exhalation phase isometric and isotonic muscle tensing occur. While the patient is breathing, the therapist should observe the posture and movement of the thoracic cage and diaphragm. Basic posture correction in sitting and walking and Sensorimotor training by the ball will be applied
  Arms: schroth exercise
Other: postural correction exercise — the patients will receive postural correction exercises, stretches, and exercises to the pectoralis major, elevator scapulae, upper trapezius, serratus anterior, rhomboids, and deep neck flexors. The stretches included sitting chair stretches, Brugger's, wall angels, and doorway stretches. The exercises included push up- plus, head-neck-retraction, and Kibler squeeze

SUMMARY:
The study will be conducted to investigate the effect of Schroth method on balance in patients with the upper cross syndrome

DETAILED DESCRIPTION:
Upper crossed syndrome (UCS) is the most common postural dysfunction in the musculature of the shoulder girdle /cervicothoracic region, which creates joint dysfunction, particularly at the atlanto-occipital joint, cervicothoracic joint C4-C5 segment, glenohumeral joint and T4-T5 segment.

The Schroth method helps patients to halt curve progression, reverse abnormal curves, reduce pain, increase vital capacity and improve posture and appearance The Schroth method consists of sensorimotor, postural, and breathing exercises aimed at recalibration of normal postural alignment, static and dynamic postural control and spinal stability.

There are no studies on Schroth method on the upper cross syndrome, so this study will be conducted to know the effective method of treatment for upper cross syndrome.. forty patients with the upper cross syndrome will be allocated randomly to two equal groups; one experimental group will receive Schroth method twice a week for four weeks and control group will receive postural correction exercise twice a week for four weeks.

ELIGIBILITY:
Inclusion Criteria:

* The patient's age ranged from 17 to 22 years
* Body mass index between 20-25 kg/m2
* The participants are diagnosed with upper cross syndrome
* Patients with normal cognitive aspects willing and able to participate in a program safely

Exclusion Criteria:

* The participants have experienced any recent trauma (within 3 months of the initial consultation)
* The participant's primary complaint is that of headaches or facial pain.
* Participants have any sort of structural abnormality in upper and middle back e.g., Scoliosis, or had a positive Adams test.
* Participants who are taking anti-inflammatory or muscle relaxant medication had to have a three-day "wash out" period before participating in the study

Ages: 17 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
stability index | up to four weeks
  stability index will be measured by Biodex balance system
spinal curvature | up to four weeks
  spinal mouse will be used to assess thoracic spine curvature. Total angle of the thoracic spine is 41-44 degree

SECONDARY OUTCOMES:
craniovertebral angle | up to four weeks
  craniovertebral angle will be measured by photogrammetric method
pain intensity | up to four weeks
  pain will be measured by visual analogue scale. It consists of a line of 10 cm with opposite edges; one edge has no pain and the other edge has the worst pain
neck function | up to four weeks
  neck function will be measured by Arabic neck disability index.. It consisting of 10 items with six choices. There is no disability for scores from 0 to 4; 5-14 is mild; 15-24 is moderate; 25-34 is severe, and finally more than 34 is a complete disability
Respiratory pulmonary functions | up to four weeks
  Respiratory pulmonary functions will be assessed by spirometry. assess breathing and respiratory ability by forced vital capacity test (FVC) and forced expiratory volume at one second test (FEV1)
shoulder posture | up to four weeks
  The shoulder's rounded position will be measured by tap measurement. the patients will be in supine and the therapist measure the distance from their shoulder to the plinth using tape measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy Cairo university, Giza, Egypt